CLINICAL TRIAL: NCT01175421
Title: Development and Validation of a Multidimensional System as Predictor of Outcomes in Obstructive Sleep Apnea: The OSA-SCORE
Brief Title: Multidimensional System as Predictor of Outcomes in Obstructive Sleep Apnea: The OSA-SCORE
Acronym: OSA-SCORE
Status: Completed | Type: Observational
Sponsor: Hospital Miguel Servet (Other)
Responsible Party: Principal Investigator, Jose M. Marin, M.D., Hospital Miguel Servet
Other Study IDs: PS09/02449
Record Dates: First submitted 2010-08-03; First posted 2010-08-04 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2010-08

CONDITIONS: Snoring; Sleep Apnea
Keywords: snoring; sleep apnea; sleep study; cardiovascular outcomes
MeSH Terms: conditions — Snoring; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing sleep study

SUMMARY:
Purpose:

In a retrospective cohort the investigators will validate, the goodness of a multidimensional index to classified the severity of patients with sleep disordered breathing that has been previously developed in a prospective longitudinal cohort.

DETAILED DESCRIPTION:
Methods. In the developing study, three variables were found as predictors of mayor outcomes and were incorporated in a multidimensional index: the apnea-hypopnea index, the severity of daytime sleepiness as quantified by the Epworth questionnaire and the presence of current cardiovascular disease. The index (OSA-SCORE) has a value between 0 (less risk) to 5 (more risk). For each point, a significant increment in the risk of death was found. In the retrospective validation study, a number of potential variables will be recorded, all of them also predictors of major outcomes. Data will be recorded by trained personnel on-site at the respiratory Sleep Units around the country. The final cohort will include 1100 subjects aged > 18 years . The observation time will be considered since the time at diagnosis to fatal event and the patient will be censored when non-invasive ventilation was started or at the recorded time if the patient is alive. The primary outcome is all-cause death.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients (> 18 years)

Exclusion Criteria:

* Under 18 years old
* Unable to complete sleep study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sleep Clinic
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2010-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
All cause mortality | Five years

SECONDARY OUTCOMES:
Cardiovascular events | Five years

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Marin, M.D., Principal Investigator — Hospital Miguel Servet
Locations (1):
- Hospital Universitario Miguel Servet, Zaragoza, Spain